CLINICAL TRIAL: NCT00465998
Title: Prediction of Labor and Delivery With the Use of Ultrasound in Pregnancies With Induced Labor
Brief Title: Study of Ultrasound Imaging to Predict Time and Outcome in Pregnancies With Induced Labor
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Norwegian University of Science and Technology (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: StaHF483201; Helse Vest 911314
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Results first posted 2016-07-19 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-06

CONDITIONS: Pregnancy; Labor, Induced
Keywords: Ultrasound; Induced labor; Cervical length; Engagement of fetal head; Occiput posterior; Outcome of labor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study was to evaluate any possible associations between engagement and position of the fetal head and the outcome of labor in women with induced labor, and to compare the value of ultrasound measurements in predicting the time from induction to delivery and operative deliveries.

DETAILED DESCRIPTION:
Fetal head engagement measured by ultrasound as a predictive factor of labor outcome in women with induced labor

T. EGGEBØ, L. K. GJESSING, I. ØKLAND, C. HEIEN, P. ROMUNDSTAD*, K. Å. SALVESEN** Department of Obstetrics and Gynaecology, Stavanger University Hospital, Norway * Department of Public Health, NTNU, Norway, St Olavs Hospital, Trondheim University Hospital

** National Center for Fetal Medicine, Department of Obstetrics and Gynaecology, Trondheim University Hospital (St. Olav's Hospital) and Department of Laboratory Medicine, Children's and Women's Health, Norwegian University of Science and Technology

KEYWORDS:

Ultrasound, induced labor, cervical length, engagement of fetal head, occiput posterior, Bishop score, outcome of labor

Objective The aim of the study is to evaluate any possible associations between engagement of the fetal head, the cervical status or occiput posterior position and the outcome of labor in women with induced labor, and to compare the value of ultrasound measurements with Bishop score in predicting operative deliveries.

Methods The ultrasound examinations will be carried out in 275 women immediately before induction of labor. A transabdominal scan will be performed to determine the position of the fetal occiput, a transperineal scan with transverse view to determine the degree of engagement and a transvaginal examination to evaluate the cervical length and the cervical angle.. The Bishop score will be performed by another examinator who is blinded to the results of the ultrasound examinations. The time from induction to delivery will be tested in a Cox regression analysis with fetal head engagement, cervical length and parity as possible predictive factors and maternal age, BMI, gestational age, birth weight and head circumference as possible confounders.

Inclusion and exclusion criteria:

Women were eligible for the study if they had a live singleton pregnancy with cephalic presentation and a gestational age of more than 37 completed pregnancy weeks according to a mid-trimester scan.

Statistical analysis Appropriate statistical tests for comparisons, such as Mann Whitney U test, chi-square test, Fisher's exact test, Pearson correlation, Kaplan Meier survival analysis and Cox regression analysis will be used. For receiver-operating characteristics (ROC) curves, the area under the curve will be used as discriminator. P-values < 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* Indication of induced labor

Exclusion Criteria:

* More than one fetus
* Less than 37 weeks of pregnancy
* Previous cesarean section
* Breach position
* Dead fetus

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant females with indication for induced labor
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2006-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Å. Salvesen, Prof. PhD, Study Director — St. Olavs Hospital
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

REFERENCES:
- [Background] BISHOP EH. PELVIC SCORING FOR ELECTIVE INDUCTION. Obstet Gynecol. 1964 Aug;24:266-8. No abstract available. PMID 14199536
- [Background] Rane SM, Guirgis RR, Higgins B, Nicolaides KH. The value of ultrasound in the prediction of successful induction of labor. Ultrasound Obstet Gynecol. 2004 Oct;24(5):538-49. doi: 10.1002/uog.1100. PMID 15386612
- [Background] Dietz HP, Lanzarone V, Simpson JM. Predicting operative delivery. Ultrasound Obstet Gynecol. 2006 Apr;27(4):409-15. doi: 10.1002/uog.2731. PMID 16565982
- [Background] Eggebo TM, Gjessing LK, Heien C, Smedvig E, Okland I, Romundstad P, Salvesen KA. Prediction of labor and delivery by transperineal ultrasound in pregnancies with prelabor rupture of membranes at term. Ultrasound Obstet Gynecol. 2006 Apr;27(4):387-91. doi: 10.1002/uog.2744. PMID 16565994
- [Background] Eggebo TM, Okland I, Heien C, Gjessing LK, Romundstad P, Salvesen KA. Can ultrasound measurements replace digitally assessed elements of the Bishop score? Acta Obstet Gynecol Scand. 2009;88(3):325-31. doi: 10.1080/00016340902730417. PMID 19172418
- [Background] Eggebo TM, Heien C, Okland I, Gjessing LK, Romundstad P, Salvesen KA. Ultrasound assessment of fetal head-perineum distance before induction of labor. Ultrasound Obstet Gynecol. 2008 Aug;32(2):199-204. doi: 10.1002/uog.5360. PMID 18528923

RESULTS

PARTICIPANT FLOW:
Groups:
- Successful Vaginal Delivery: 275 women with induced labors were included in the study, and the main outcome was vaginal delivery.
  Variables associated to a successful vaginal delivery was examined.
Period: Overall Study
Arm/Group | Successful Vaginal Delivery
Started | 275
Completed | 275
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Time From Induction to Delivery: Variables associated to time from induction to delivery were investigated.
Arm/Group | Time From Induction to Delivery
Number analyzed (Participants) | 275
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 272
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 30 [18 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275
  Male | 0
Region of Enrollment [Number; unit: participants]
  Norway | 275

OUTCOME MEASURES:

1. Primary Outcome: Vaginal Delivery in Induced Labors
Description: The association between Bishop score, ultrasound assessed fetal station, ultrasound assessed cervical length, cervical posterior angle and a vaginal delivery was investigated using area under the ROC curves. Fetal station was assessed by ultrasound as the fetal head-perineum distance (HPD); which was measured by transperineal ultrasound imaging as the shortest distance from the outer bony limit of the fetal skull to the skin surface of the perineum.
Time Frame: Time from induction of labor to delivery
Measure: Number (95% Confidence Interval); unit: percentage of area under the ROC curve
Arm/Group | Successful Vaginal Delivery
Number analyzed (Participants) | 275
percentage of area under the ROC curve
  Area under the ROC curve associated to HPD | 62 [52 to 71]
  Area under the curve associated to cervical length | 61 [51 to 71]
  Area under the curve associated to cervical angle | 63 [52 to 74]
  Area under the curve associated to Bishop score | 60 [51 to 69]

2. Secondary Outcome: Delivery Within 24 Hours
Description: Association between parity, HPD, cervical length, cervical angle, occiput posterior position, parity, BMI and the Hazard ratio of delivering within 24 hours was investigated using Cox regression analysis.
Time Frame: Time from induction to delivery
Population: Hazard ratio was reported.
Measure: Number (95% Confidence Interval); unit: Hazard ratio
Arm/Group | Time From Induction to Delivery
Number analyzed (Participants) | 275
Hazard ratio
  HPD ≤ 40 mm | 1.67 [1.23 to 2.26]
  Cervical length ≤ 25 mm | 2.35 [1.75 to 3.14]
  Cervical posterior > 90 degrees | 1.92 [1.22 to 3.04]
  Occiput posterior position | 1.27 [0.93 to 1.75]
  Multiparous woman | 3.25 [2.43 to 4.35]
  BMI < 30 | 1.14 [0.78 to 1.65]

ADVERSE EVENTS:
Time Frame: From start of induction to discharge from the labor ward
Arm/Group | Successful Vaginal Delivery
Serious Adverse Events (participants affected / at risk) | 1/275
Other Adverse Events (participants affected / at risk) | 0/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Successful Vaginal Delivery (N=275)
maternal death (Cardiac disorders) | 1 (1) — One woman had a sudden cardiac arrest 10 h after induction of labor due to amniotic fluid embolism. A healthy baby was delivered, but the mother died. An investigation concluded that the event was not associated to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes